CLINICAL TRIAL: NCT01702324
Title: Evaluation of DD-25 Topical Cream for the Treatment of Psoriasis Vulgaris : Proof of Concept Study
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fortuderm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DD-25; 0290-12-TLV (Other: Tel Aviv Sourasky Medical Center)
Record Dates: First submitted 2012-10-03; First posted 2012-10-08 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Psoriasis Vulgaris
Keywords: Psoriasis Vulgaris; Plaque; Topical; Treatment
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DD-25 (Experimental): A concentration of 0.025% of topical DD-25 cream.
  Interventions: Drug: DD-25

INTERVENTIONS:
Drug: DD-25 — A topical DD-25 cream at 0.025% concentration.
  Other Names: Fortuderm DD-25 Psoriasis Cream

SUMMARY:
The purpose of this study is to determine the efficacy of DD-25, a new topical drug, on plaque Psoriasis Vulgaris.

The study will include subjects at plaque stage from 5-20% body area involvement. A total of 30 subjects will be treated with cream application on affected areas twice daily for three weeks.The efficacy of the preparation will be documented by PASI score, Global physician assessment and photos.

DETAILED DESCRIPTION:
Psoriasis Vulgaris remains a widespread clinical entity with chronic outflares and various regimens of treatment, none of them definitive. A new safe and efficacious, external treatment is required for.

ELIGIBILITY:
Inclusion Criteria:

1. Subject age 18-60
2. Diagnosis of PS by a dermatologist with lesions on arms, legs or trunk
3. Subjects have stable plaque PS, mild to moderate form, Body Surface Area of 5-20%.
4. Subject understood and signed an informed consent form

Exclusion Criteria:

1. Guttate, erythrodermic, palm-plantar or pustular psoriasis as sole or predominant form of psoriasis.
2. Hypersensitivity to sunlight; history of Lupus, PMLE, or any disease known to be worsened by UV light exposure
3. Pregnancy, breast feeding
4. History of cancer, excluding non-melanoma skin cancer.
5. Patients with history of ischemic heart disease (e.g. angina pectoris, myocardial infarction); cerebrovascular syndromes, peripheral vascular or uncontrolled hypertension. Subjects with known severe hepatic and/or severe renal insufficiency.
6. Any medical condition that, in the opinion of the Investigator, would jeopardize the health of the patient during the course of this study.
7. Systemic treatment with biological therapies with a possible effect on psoriasis vulgaris within 4 months or 5 drug half-lives prior to checkup.
8. Systemic treatments with all other therapies than biologicals, with a potential effect on psoriasis vulgaris (e.g., corticosteroids, vitamin D analogues, retinoids, immuno-suppressants) within the 8-week period prior to randomization. Subjects using within the 8 week period prior to randomization PUVA or Phototherapy. Use of SSRI or MAO inhibitors.
9. Subjects using one of the following TOPICAL drugs for the treatment of PS within 2 weeks prior to randomization: e.g. WHO group I-II corticosteroids, retinoids, Vit. D analogues, immunomodulators, Anthracene derivatives, Salicylic acid.
10. Subjects with current participation in any other interventional clinical or subjects with any concomitant dermatological disorder(s) which might preclude accurate evaluation of the psoriasis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy after 3 weeks as compared to baseline. | 3 weeks
  Evaluation of the effectiveness of DD-25 over a period of 3 weeks treatment by analyzing the changes in the Psoriasis Area & Severity Index (PASI) in moderate to mild Plaque Psoriasis patients. Improvement to be assessed by changes in erythema, induration and desquamation as seen on days 0, 10 and 21.

SECONDARY OUTCOMES:
PASI reduction of 50% | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hagit Matz, M.D., Principal Investigator — Dept of Dermatology, Tel Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Tel Aviv, Israel